CLINICAL TRIAL: NCT02512055
Title: Ketamine Tolerance in Children After Repeated Administrations During Radiotherapy Sessions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Oya Yalcin Cok, Associate Professor, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KA09/247
Record Dates: First submitted 2015-07-24; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Conscious Sedation Failure During Procedure
MeSH Terms: interventions — Ketamine; Atropine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental): Pediatric patients undergoing repeat radiotherapy session under ketamine sedation
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Repeated ketamine 2 mg/kg administration intravenously for sedation during each radiotherapy sessions
  Other Names: Atropine

SUMMARY:
Ketamine provides a safety zone for sedated but spontaneously ventilated children especially in remote conditions such as radiotherapy units where sedation is an essential practice for children to keep calm and motionless In this study, investigators planned to analyse ketamine doses needed and the recovery times in pediatric oncology patients undergoing repeated radiotherapy sessions.

DETAILED DESCRIPTION:
Ketamine provides a safety zone for sedated but spontaneously ventilated children especially in remote conditions such as radiotherapy units where sedation is an essential practice for children to keep calm and motionless.However, there had been a disagreement about the ketamine doses needed for a continuous and steady level of sedation during repeated radiotherapy sessions in children. In this study, investigators planned to analyse ketamine doses needed and the recovery times in pediatric oncology patients undergoing repeated radiotherapy sessions.After approval from the Baskent University, School of Medicine, Ethics and Research Committee (KA09/247) and informed consents of the patients' guardians, 33 pediatric patients undergoing radiotherapy due to oncologic disorders were enrolled to receive ketamine 2 mg/kg and atropine 10 μg/kg.Patients' demographic data such as age, gender, weight, ASA physical status and duration and total number of radiotherapy sessions were noted. Total ketamine consumption to maintain the targeted sedation level during each session, additional dose administration and the recovery time were recorded. The adverse events such as apnea, laryngospasm, bronchospasm, desaturation, respiratory depression, bradycardia, sedation levels deeper or superficial than intended to, excessive salivation, allergy, nausea and vomiting and need for emergency medication were also noted after each session. The study drugs were prepared, labelled and administered by an anesthetist according to the study protocol and data were recorded by an anesthetist blind to the amount of the study drug used.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing radiotherapy due to oncologic disorders

Exclusion Criteria:

* Patients younger than 1 year and older than 14 year,
* patients with cardiac, renal or liver function abnormalities, who were already under sedative drug treatment or allergic to the drugs to be used or the patients for whom the study drugs

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Total ketamine consumption during each session | peroperative 3 hours

SECONDARY OUTCOMES:
Recovery time | peroperative 3 hours

REFERENCES:
- [Background] Hoffman GM, Nowakowski R, Troshynski TJ, Berens RJ, Weisman SJ. Risk reduction in pediatric procedural sedation by application of an American Academy of Pediatrics/American Society of Anesthesiologists process model. Pediatrics. 2002 Feb;109(2):236-43. doi: 10.1542/peds.109.2.236. PMID 11826201
- [Background] Lois F, De Kock M. Something new about ketamine for pediatric anesthesia? Curr Opin Anaesthesiol. 2008 Jun;21(3):340-4. doi: 10.1097/ACO.0b013e3282f82bde. PMID 18458551
- [Background] Macnab AJ, Levine M, Glick N, Susak L, Baker-Brown G. A research tool for measurement of recovery from sedation: the Vancouver Sedative Recovery Scale. J Pediatr Surg. 1991 Nov;26(11):1263-7. doi: 10.1016/0022-3468(91)90594-j. PMID 1812252
- [Background] Tobias JD. Tolerance, withdrawal, and physical dependency after long-term sedation and analgesia of children in the pediatric intensive care unit. Crit Care Med. 2000 Jun;28(6):2122-32. doi: 10.1097/00003246-200006000-00079. PMID 10890677
- [Background] Trujillo KA, Akil H. Inhibition of opiate tolerance by non-competitive N-methyl-D-aspartate receptor antagonists. Brain Res. 1994 Jan 7;633(1-2):178-88. doi: 10.1016/0006-8993(94)91538-5. PMID 8137155
- [Background] Trujillo KA. The neurobiology of opiate tolerance, dependence and sensitization: mechanisms of NMDA receptor-dependent synaptic plasticity. Neurotox Res. 2002 Jun;4(4):373-91. doi: 10.1080/10298420290023954. PMID 12829426
- [Background] Trujillo KA, Zamora JJ, Warmoth KP. Increased response to ketamine following treatment at long intervals: implications for intermittent use. Biol Psychiatry. 2008 Jan 15;63(2):178-83. doi: 10.1016/j.biopsych.2007.02.014. Epub 2007 Jun 13. PMID 17568566
- [Background] Zapantis A, Leung S. Tolerance and withdrawal issues with sedation. Crit Care Nurs Clin North Am. 2005 Sep;17(3):211-23. doi: 10.1016/j.ccell.2005.04.011. PMID 16115529